CLINICAL TRIAL: NCT06396936
Title: Investigation of the Effects of Physical Activity on Smartphone Addiction, Pain and Sleep Quality in Young Adults
Brief Title: The Effect of Calisthenic Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KTOKARACA002
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-04

CONDITIONS: Physical Inactivity; Sleep Hygiene; Smartphone Addiction; Pain
Keywords: Physical Inactivity; Sleep Hygiene; Smartphone Addiction; Pain
MeSH Terms: conditions — Sedentary Behavior; Sleep Hygiene; Internet Addiction Disorder; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Calisthenic exercise program
  Interventions: Other: Calisthenic exercise program
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Other: Calisthenic exercise program — Calisthenic exercises to be applied in our study; These are exercises that are performed by creating resistance only with your body weight, without the need for any equipment or gym.
  Arms: Study Group

SUMMARY:
This study will investigate the effects of physical activity in young adults. With the increase in physical activity, the change in smartphone addiction, pain and sleep quality parameters will be evaluated.

DETAILED DESCRIPTION:
This study aims to increase physical activity with a calisthenic exercise program. An answer will be sought to the question of whether increased physical activity causes changes in phone addiction, pain and sleep quality parameters.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study.
* Being between the ages of 15-35.

Exclusion Criteria:

* Individuals with an orthopedic and/or neurological disease that will affect their sleep health and/or pain level,
* Individuals with physical disabilities,
* Individuals who have undergone any surgical procedure in the last 6 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | The evaluation will be applied at the beginning of the treatment program.
  Pittsburgh Sleep Quality Index will used to evaluate overall sleep quality in young adults.
Smartphone addiction | The evaluation will be applied at the beginning of the treatment program.
  The short version of the smartphone addiction scale (SAS-SV) will used to evaluate smartphone addiction.
Physical Activity | The evaluation will be applied at the beginning of the treatment program.
  The International Physical Activity Survey will used to evaluate physical activity.
Levels of Quality of life | The evaluation will be applied at the beginning of the treatment program.
  Short Form Health Survey (SF-36) will used to evaluate health status.

SECONDARY OUTCOMES:
Pain intensity (neck pain and head pain) | The evaluation will be applied at the beginning of the treatment program
  The Visual Analogue Scale (VAS) will used to measure pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Osman Karaca, PhD, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not sharing other researchers.